CLINICAL TRIAL: NCT07202949
Title: EAT-UP - Extended Antibiotic Treatment in Chronic UTI Patients; a Phase II Safety and Efficacy Trial
Brief Title: A Clinical Trial of Extended (High) Treatment Dose Antibiotics in Combination With Methenamine Hippurate Compared to the Standard of Care (Either Prophylactic (Low) Dose Antibiotic Treatment or Methenamine Hippurate) in Females With Chronic Urinary Tract Infection
Acronym: EAT-UP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 155876; CTU/2019-342 (Other: Comprehensive Clinical Trial Unit, UCL)
Record Dates: First submitted 2025-09-16; First posted 2025-10-02 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Urinary Tract Infection
Keywords: Urinary Tract Infection; Antibiotics; Urological Diseases; methenamine hippurate; Cefalexin; Nitrofurantoin; Trimethoprim; Amoxicillin; Chronic Urinary Tract Infection; UTI
MeSH Terms: conditions — Urinary Tract Infections; Urologic Diseases | interventions — methenamine hippurate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment dose antibiotic in combination with methenamine hippurate (Experimental)
  Interventions: Drug: Treatment dose antibiotic in combination with methenamine hippurate
- Prophylactic dose antibiotic or methenamine hippurate monotherapy (Active Comparator)
  Interventions: Drug: Prophylactic dose antibiotic or methenamine hippurate monotherapy

INTERVENTIONS:
Drug: Treatment dose antibiotic in combination with methenamine hippurate — Arm A includes treatment with one of three treatment dose antibiotic options, selected by the treating clinician, in combination with methenamine hippurate. Participants allocated to this arm will receive combination therapy, consisting of one of the following antibiotics:
  * Cefalexin (500mg four times daily), or
  * Nitrofurantoin (100mg twice daily), or
  * Trimethoprim (200mg twice daily) in combination with Methenamine Hippurate (1g twice daily) for 12 weeks.
  Arms: Treatment dose antibiotic in combination with methenamine hippurate
Drug: Prophylactic dose antibiotic or methenamine hippurate monotherapy — Arm B includes treatment with one of four prophylactic dose antibiotics or methenamine hippurate, but not both, selected by the treating clinician. Participants in this arm will receive monotherapy of one of the following:
  * Amoxicillin (250mg once daily), or
  * Cefalexin (125mg once daily), or
  * Nitrofurantoin (50mg once daily), or
  * Trimethoprim (100mg once daily), or
  * Methenamine Hippurate (1g twice daily) for 12 weeks.
  Arms: Prophylactic dose antibiotic or methenamine hippurate monotherapy

SUMMARY:
Chronic Urinary Tract Infection (UTI) is a type of UTI where symptoms are constant and occur every day, unlike recurrent UTIs, which come and go with symptom-free breaks in between. Current treatment for chronic UTI within the NHS is based on recommended guidelines for recurrent UTI. The standard approach typically includes one of the following treatments:

* Long-term, prophylactic (low) dose daily antibiotic (where medication is used at low doses to try to prevent symptoms reoccurring).
* Long-term use of a urinary antiseptic (which helps keep your urine bacteria free), called methenamine hippurate.

These often do not work for people with chronic UTI, and symptoms can persist. Moreover, standard urine tests may fail to detect infections, making diagnosis and treatment more challenging.

The EAT-UP trial will investigate whether longer courses of treatment (higher) dose antibiotics combined with methenamine hippurate (a urinary antiseptic) are a more effective treatment at reducing levels of infection and symptoms than standard of care treatments (as described above).

DETAILED DESCRIPTION:
EAT-UP is a UK multi-centre, randomised, open label, parallel-group, superiority, interventional phase II trial, aiming to recruit 192 female participants. Participants will undergo screening to evaluate their eligibility to participate in the trial. If eligible, participants will be randomly assigned into one of two groups:

Group 1 will receive a treatment dose antibiotic in combination with the urinary antiseptic, methenamine hippurate (1 g twice daily). The treating clinician will select one of the following antibiotics based on the individual needs of the participant, such as their medical history, concomitant medications and any known allergies:

* Cefalexin (500mg four times daily), or
* Nitrofurantoin (100mg twice daily), or
* Trimethoprim (200mg twice daily)

Group 2 will receive a low-dose prophylactic antibiotic or the urinary antiseptic, methenamine hippurate. The treating clinician will select one of the following treatments based on the individual needs of the participant, such as their medical history, concomitant medications and any known allergies:

* Amoxicillin (250mg once daily), or
* Cefalexin (125mg once daily), or
* Nitrofurantoin (50mg once daily), or
* Trimethoprim (100mg once daily), or
* Methenamine Hippurate (1g twice daily)

Participants will be taking trial medication for 12 weeks and will be required to attend clinic for assessments every 4 weeks. Participant will complete questionnaires and provide blood, urine, and perineal (the area between the vagina and anus) swabs samples.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of chronic UTI, without structural or functional urinary tract abnormality*, defined as daily persistent symptoms affecting storage (urinary frequency, urgency or urge incontinence) and urinary tract pain symptoms (including bladder pain, urethral pain, or dysuria), for at least 3 months prior to the screening visit, with previously associated transient symptomatic improvement to antibiotic treatment for UTI, which in the opinion of the delegated clinician is secondary to chronic urinary tract infection.
2. A fresh urine microscopy examination showing ≥20 white blood cells/µl of urine at the screening visit.
3. Female** patients.
4. Aged ≥18 years.
5. Screening blood result of eGFR ≥45ml/min/1.73m2.
6. Able and willing to attend trial visits and comply with all study procedures for the duration of the trial.
7. Able and willing to provide informed consent prior to any study related assessments and/or procedures.

   * A structural or functional abnormality may include kidney reflux, current or long-term catheter use, renal transplant, diversion surgery, renal stones, grade 2 or above utero-vaginal prolapse or incomplete bladder emptying.

     * For the purposes of this trial, a female will be defined as an individual assigned female at birth who has a female urinary tract.

Exclusion Criteria:

1. Inability to take at least one of the following antibiotics: Cefalexin, Nitrofurantoin, or Trimethoprim, at prophylactic and treatment dose according to NICE guidelines, and/or the Summary of Product Characteristics (such as hepatic or renal dysfunction), or any other medical contraindications.
2. Inability to take methenamine hippurate due to medical contraindications.
3. Current use of immune-modulating drugs for the treatment of chronic illnesses such as rheumatoid arthritis, chronic lung disease, any other autoimmune conditions or cancer.
4. Current use of Sodium-Glucose Transport Protein 2 (SGLT2) inhibitors*.
5. A current diagnosis of bladder cancer.
6. A diagnosis of an active sexually transmitted infection or a recent diagnosis of a sexually transmitted infection within the last 3 months of the screening visit.
7. Previous use of an antibiotic at treatment dose as per NICE guidelines for more than 14 consecutive days for treatment of UTI in the last 3 months prior to the screening visit.
8. Pregnancy (or planned pregnancy during trial participation) and/or breastfeeding.
9. Women of childbearing potential that are unable/unwilling to use an acceptable method of contraception (as described in section 3.4.1) to avoid pregnancy for the duration of the trial and for 1 week after the last dose of trial medication.
10. Current participation in another clinical trial of a device, interventional medicinal product, advanced therapy, or surgical procedure; or previous participation within 6 months of the screening visit.
11. Any medical condition or previous treatment which in the investigator's opinion compromises the potential participant's ability to participate.

    * Patient's must not have taken a Sodium-Glucose Transport Protein 2 (SGLT2) inhibitor within 24 hours before the screening visits to be eligible for the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in urinary white blood cell (WBC) count from baseline to Week 12. | Baseline, Week 4, Week 8, Week 12
  Urinary white blood cell (WBC) count, measured using fresh urine microscopy, will be used as the principal biomarker to indicate urinary tract inflammation.

SECONDARY OUTCOMES:
Changes in EuroQol EQ-5D 5-Level Health Related Quality of Life Questionnaire (EQ-5D-5L) scores at week 12, adjusted for baseline | Baseline, Week 12
  The EQ-5D-5L is a participant self-reported questionnaire which evaluates the generic quality of life at the time of completion. It comprises of a 5 item questionnaire (assessing - mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and a visual analogue scale (VAS). Each dimension assessed has 5 response scales to select from: no problems, slight problems, moderate problems, severe problems, and extreme problems
Changes in ICIQ Lower Urinary Tract Symptoms quality of life (ICIQ-LUTSqol) | Baseline, Week 4, Week 8, Week 12
  The ICIQ Lower Urinary Tract Symptoms Quality of Life (ICIQ-LUTSqol) is designed to assess the impact of lower urinary tract symptoms (LUTS) on a patient's quality of life. It consists of 19 items that explore various aspects of daily living affected by LUTS, including physical, social, emotional, and psychological domains. Responses are measured using a Likert scale, allowing clinicians and researchers to quantify the burden of symptoms and evaluate changes over time.
Changes in Whittington 39-point Lower Urinary Tract Symptoms (W-39 LUTS) scores at week 12, adjusted for baseline | Baseline, Week 4, Week 8, Week 12
  The Whittington 39-point Lower Urinary Tract Symptoms (W-39 LUTS) is a questionnaire designed to assess participant's experiences of lower urinary tract symptoms (LUTS). It consists of 39 items that explore the following LUTS symptom groups: Urgency, Pain, Stress Incontinence and Voiding.
Patient Global Impression of Improvement (PGI-I) scores at week 12. | Week 4, Week 8, Week 12
  The Patient Global Impression of Improvement (PGI-I) is used to assess a participant's perception of change in their condition following treatment. It consists of a single-item questionnaire where patients rate their overall improvement on a 7-point Likert scale, ranging from "very much better" to "very much worse."
Participant satisfaction with medication using Lübeck Medication Satisfaction (LMS) Questionnaire scores at week 12 | Week 12
  The Lübeck Medication Satisfaction (LMS) Questionnaire is designed to assess participant satisfaction with their trial medication. It comprises 18 items that evaluate satisfaction across domains such as effectiveness, side effects, ease of use, and overall contentment.
Treatment adherence assessed by the MARS-5 questionnaire at weeks 4, 8 and 12. | Week 4, Week 8 and Week 12
  The Medication Adherence Report Scale (MARS-5) is a self-report questionnaire used to assess medication adherence behaviour in participants with chronic conditions. It includes 5 items that measure both intentional and unintentional non-adherence, such as forgetting to take medication or altering doses. Each item is rated on a 5-point Likert scale, with higher scores indicating better adherence.
Frequency of rescue therapy use for participants requiring further treatment escalation for an acute flare of symptoms at 12 | Week 4, Week 8 and Week 12
  Participants will be prescribed rescue therapies, typically short courses of antibiotics at higher doses than their assigned treatment arm, in response to acute symptom flares. The use and effectiveness of these therapies will be reviewed at each trial visit.
Changes in urine culture species, cfu/ml count, sensitivities and resistance profiles at week 12, adjusted for baseline | Baseline and Week 12
  Urine samples will be submitted to the central laboratory for testing to evaluate the changes in the type of bacteria found in the urine, the amount of bacteria and how the bacteria is responding to antibiotics (including resistance).
Changes in Perineal swab analyses of E.coli identified, sensitivities and resistance profiles at week 12, adjusted for baseline | Baseline and Week 12
  A swab will be taken from the area between the vagina and anus (this is called the perineal area) either by the participant (self-swab) or with assistance from the local research team. The swab will be submitted to the central laboratory for testing. The tests will be used to measure any changes in how bacteria in the gut responds to antibiotics (also known as antimicrobial resistance).
Safety and tolerability of the intervention as indicated by changes in pulse (bpm) from baseline to Week 12 | Baseline, Week 4, Week 8 and Week 12
  Vital signs
Safety and tolerability of the intervention as indicated by changes in blood pressure (mmHg) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Vital signs
Safety and tolerability of the intervention as indicated by changes in temperature (°) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Vital signs
Safety and tolerability of the intervention as indicated by changes in respiratory rate (breaths per minute)from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Vital signs
Safety and tolerability of the intervention as indicated by changes in weight (kg) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Vital signs
Safety and tolerability of the intervention as indicated by changes in Haemoglobin (g/dL) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Full Blood Count)
Safety and tolerability of the intervention as indicated by changes in Red Blood Cell Count (10^12/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Full Blood Count)
Safety and tolerability of the intervention as indicated by changes in Platelets (10^9/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Full Blood Count)
Safety and tolerability of the intervention as indicated by changes in total White Blood Cell Count (10^9/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Full Blood Count)
Safety and tolerability of the intervention as indicated by changes in Neutrophils (10^9/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Full Blood Count)
Safety and tolerability of the intervention as indicated by changes in Lymphocytes (10^9/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Full Blood Count)
Safety and tolerability of the intervention as indicated by changes in Monocytes (10^9/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Full Blood Count)
Safety and tolerability of the intervention as indicated by changes in Eosinophils (10^9/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Full Blood Count)
Safety and tolerability of the intervention as indicated by changes in Basophils (10^9/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Full Blood Count)
Safety and tolerability of the intervention as indicated by changes in Albumin (g/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Biochemistry)
Safety and tolerability of the intervention as indicated by changes in Total Bilirubin (µmol/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Biochemistry)
Safety and tolerability of the intervention as indicated by changes in Alanine Transaminase (ALT) (IU/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Biochemistry)
Safety and tolerability of the intervention as indicated by changes in Alkaline Phosphatase (ALP) (IU/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Biochemistry)
Safety and tolerability of the intervention as indicated by changes in Calcium (mmol/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Biochemistry)
Safety and tolerability of the intervention as indicated by changes in Carbon dioxide (bicarbonate) (mmol/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Biochemistry)
Safety and tolerability of the intervention as indicated by changes in Chloride (mmol/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Biochemistry)
Safety and tolerability of the intervention as indicated by changes in Creatinine (µmol/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Biochemistry)
Safety and tolerability of the intervention as indicated by changes in Estimated Glomerular Filtration Rate (eGFR) (ml/min/1.72m²) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Biochemistry)
Safety and tolerability of the intervention as indicated by changes in Glucose (mmol/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Biochemistry)
Safety and tolerability of the intervention as indicated by changes in Phosphorus inorganic (phosphate) (mmol/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Biochemistry)
Safety and tolerability of the intervention as indicated by changes in Potassium (mmol/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Biochemistry)
Safety and tolerability of the intervention as indicated by changes in Sodium (mmol/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Biochemistry)
Safety and tolerability of the intervention as indicated by changes in Urea (mmol/L) from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Standard diagnostic laboratory test (Biochemistry)
Safety and tolerability of the intervention as indicated by the occurrence / severity of treatment related Adverse Events assessed by CTCAE v5.0 from baseline to week 12 | Baseline, Week 4, Week 8 and Week 12
  Number of participants with treatment related adverse events assessed by CTCAE v5.0 from baseline to week 12

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Whittington Health NHS Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Undecided